CLINICAL TRIAL: NCT07312721
Title: Comparative Effectiveness of Triple Versus Quadruple Therapy in the Treatment of Helicobacter Pylori Induced Gastritis: A Randomized Controlled Trial
Brief Title: Comparative Effectiveness of Triple Versus Quadruple Therapy in the Treatment of Helicobacter Pylori Induced Gastritis
Acronym: HP-THERAPY-TRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azfar Farogh (Other)
Responsible Party: Sponsor-Investigator, Azfar Farogh, Professor of Medicine, Shahida Islam Medical Complex
Organization: Shahida Islam Medical Complex (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIMC/ETC/0008/24
Record Dates: First submitted 2025-12-13; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Helicobacter Pylori Infection; Chronic Gastritis; Peptic Ulcer Disease
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triple Therapy Group (Experimental): Participants received Omeprazole 40 mg twice daily, Amoxicillin 1 g twice daily, and Clarithromycin 500 mg twice daily for 14 days.
  Interventions: Drug: Triple Therapy
- Quadruple Therapy Group (Experimental): Participants received Omeprazole 40 mg twice daily, Metronidazole 400 mg three times daily, Tetracycline 500 mg every six hours, and Bismuth subsalicylate for 14 days.
  Interventions: Drug: Quadruple Therapy

INTERVENTIONS:
Drug: Triple Therapy — Omeprazole 40 mg BID, Amoxicillin 1 g BID, Clarithromycin 500 mg BID for 14 days.
  Arms: Triple Therapy Group
Drug: Quadruple Therapy — Omeprazole 40 mg BID, Metronidazole 400 mg TID, Tetracycline 500 mg QID, Bismuth subsalicylate for 14 days.
  Arms: Quadruple Therapy Group

SUMMARY:
This randomized controlled trial is designed to compare the efficacy of standard triple therapy versus bismuth-based quadruple therapy for the eradication of Helicobacter pylori-induced gastritis. The study is being conducted at Shahida Islam Medical College, Lodhran, Pakistan. Adult patients with confirmed H. pylori infection are randomly allocated to receive either a 14-day triple therapy regimen or a 14-day bismuth-based quadruple therapy regimen. Eradication of H. pylori is assessed six weeks after completion of treatment using stool antigen testing. The primary outcome measure is the proportion of patients achieving successful eradication of H. pylori.

DETAILED DESCRIPTION:
Background:

Helicobacter pylori infection is a major cause of chronic gastritis, peptic ulcer disease, and gastric malignancy. Standard triple therapy has historically been used as first-line treatment; however, increasing antibiotic resistance has led to declining eradication rates in many regions. Bismuth-based quadruple therapy has emerged as an alternative regimen and is recommended in areas with suspected or confirmed antibiotic resistance.

Objective:

To compare the efficacy of standard triple therapy versus bismuth-based quadruple therapy in achieving eradication of Helicobacter pylori in adult patients with H. pylori-induced gastritis.

Study Design and Methods:

This is a randomized controlled trial conducted in the Department of Medicine at Shahida Islam Medical College, Lodhran, Pakistan. Adult patients aged 18 to 65 years with confirmed H. pylori infection based on stool antigen testing are eligible for inclusion. Participants are randomly assigned in a 1:1 ratio to one of two treatment groups. One group receives standard triple therapy consisting of omeprazole, amoxicillin, and clarithromycin for 14 days. The second group receives bismuth-based quadruple therapy consisting of omeprazole, metronidazole, tetracycline, and bismuth subsalicylate for 14 days.

Patients are followed for six weeks after completion of therapy. Eradication of H. pylori is evaluated using repeat stool antigen testing. The primary outcome measure is successful eradication of H. pylori. Secondary analyses include assessment of eradication outcomes across demographic and clinical subgroups.

Ethical Approval:

The study protocol has been approved by the Institutional Review Board of Shahida Islam Medical College (IRB No. SIMC/ETC/0008/24, dated 05 January 2024). Written informed consent is obtained from all participants prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.

Confirmed Helicobacter pylori infection based on a positive stool antigen test.

Willing and able to provide written informed consent.

Exclusion Criteria:

History of allergy or hypersensitivity to any of the study drugs (omeprazole, amoxicillin, clarithromycin, metronidazole, tetracycline, or bismuth compounds).

Prior H. pylori eradication therapy.

Pregnancy or lactation.

History of gastrointestinal bleeding, peptic ulcer perforation, or prior gastric surgery.

Chronic renal failure or hepatic dysfunction.

Current use of proton pump inhibitors or antibiotics within the previous six weeks.

Use of traditional (Hakeem) medications or herbal remedies affecting gastric function.

Psychiatric illness or inability to comply with treatment and follow-up.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Eradication of Helicobacter pylori infection six weeks post-treatment | 6 weeks after treatment completion
  Eradication was assessed by stool antigen testing six weeks after completion of therapy. A negative stool antigen test indicated successful eradication.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Azfar Farogh, Principal Investigator — Shahida Islam Medical College, Lodhran
Locations (1):
- Shahida Islam Medical College, Lodhran, Lodhran, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Miao R, Chen J, Gao S, Wang L, Zhou W, Wan C, Wang Z. A randomised controlled clinical study of standard triple therapy, bismuth-based quadruple therapy and sequential therapy for Helicobacter pylori infection in children. BMC Pediatr. 2024 Aug 23;24(1):543. doi: 10.1186/s12887-024-05020-6. PMID 39180014